CLINICAL TRIAL: NCT01691417
Title: The Impact of Intermittent Sequential Pneumatic Compression (ISPC) Leg Sleeves on Cardiac Performance in Patients With Congestive Heart Failure
Brief Title: Pneumatic Sleeves and Congestive Heart Failure
Acronym: Sleeves-Bickel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Sponsor
Other Study IDs: Sleeves-Bickel
Record Dates: First submitted 2012-09-09; First posted 2012-09-24 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

ARMS (2):
- Pneumatic Sleeves (Experimental)
  Interventions: Device: Intermittent Sequntial Pnumatic Compression Leg Sleeves
- Congestive Heart Failure Patients (Experimental)
  Interventions: Device: Intermittent Sequntial Pnumatic Compression Leg Sleeves

INTERVENTIONS:
Device: Intermittent Sequntial Pnumatic Compression Leg Sleeves

SUMMARY:
Based on the reversal of the adverse cardiovascular parameters during Laproscopic Surgery and its influence on cardiac activity in healthy subjects, the investigators expect to improved cardiac function in patients suffering from congestive heart failure.

ELIGIBILITY:
Inclusion Criteria:

* CHF (as clinically evaluated and asessed by TTE)
* Gave informed consent
* NYHA Class II-III
* LVEF equal or less than 40%

Exclusion Criteria:

* Patients who could not sign informed consent
* NYHA Class IV
* Oxygen saturation less than 90% under room air

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

PRIMARY OUTCOMES:
Cardiac Output

SECONDARY OUTCOMES:
Systemic vascular resistance

OTHER OUTCOMES:
Stroke volume

CONTACTS AND LOCATIONS:
Locations (1):
- Western Galilee Hospital, Nahariya, Israel